CLINICAL TRIAL: NCT04417010
Title: A Prospective Study to Identify KRAS Gene and Safe Margin in Association With Outcome in Colorectal Liver Metastases Following Ultrasound-guided Radiofrequency Ablation
Brief Title: To Identify KRAS Gene and Safe Margin in Association With Outcome in Colorectal Liver Metastases Following Ultrasound-guided Radiofrequency Ablation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Kun Yan, director, Peking University Cancer Hospital & Institute
Other Study IDs: 2020-2-2152
Record Dates: First submitted 2020-06-02; First posted 2020-06-04 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: KRAS Gene; Colorectal Cancer; Liver Metastasis; Safe Margin; Radiofrequency Ablation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Radiofrequency Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Radiofrequency ablation — Both groups of patients underwent radiofrequency ablation

SUMMARY:
To investigate the clinical effect of radiofrequency ablation on colorectal cancer liver metastases with different KRAS gene status

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed as liver metastasis of colorectal cancer;
2. There are no more than 3 liver metastases and all the lesions are not more than 5 cm; or no more than 6 liver metastases and all the lesions are not more than 3.0 cm;
3. The primary lesion of colorectal cancer has been treated curatively or is planned to undergo curative treatment;
4. KRAS gene test results can be obtained for primary or metastatic foci;
5. Signing informed consent voluntarily;
6. Men or women who have reached the age of 18;
7. Ultrasound or ultrasound contrast can clearly show the lesion and guide RFA treatment;
8. Platelet count> 50,000/mm3, prothrombin activity> 50%;
9. Child-Pugh grade A or B of liver disease, but no hepatic encephalopathy or/and ascites;
10. Subjects are willing to return to the research center for research follow-up;
11. Life expectancy ≥ 6 months-

Exclusion Criteria:

1. suffer from but not limited to the following serious diseases: congestive heart failure, myocardial infarction or cerebrovascular accident, or life-threatening arrhythmia in the past 6 months;
2. During pregnancy or lactation. Before receiving research treatment, women of childbearing age must have a negative serum pregnancy test;
3. Any known allergic reactions to the intravenous imaging agent used in this study;
4. There is portal vein or hepatic vein tumor infiltration/carcinoma;
5. International normalized ratio of prothrombin> 1.5 times the upper limit of normal value (UNL) of the research center;
6. Platelet count <50,000/mm3, absolute neutrophil count <1500/mm3, or heme value <10.0g/dL;
7. Serum creatinine ≥2.5mg/dL or calculated creatinine clearance (CrCl) ≤25.0ml/min;
8. Serum bilirubin>3.0mg/dL;
9. Serum albumin <2.8g/dL;
10. Body temperature >101°F (38.3°C) immediately before study treatment;
11. being treated with other research drugs;
12. Heart failure NYHA function grade is III or IV .

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Men or women 18 years of age or older
Sampling Method: Probability Sample
Enrollment: 163 (Estimated)
Dates: Start 2020-06-01 (Estimated); Primary Completion 2023-05-31 (Estimated); Study Completion 2023-05-31 (Estimated)

PRIMARY OUTCOMES:
local tumor progression | 2020-06-01-2023-05-31
  the appearance of tumor foci at the edge of the ablation zones after at least one contrast-enhanced follow-up study has documented adequate ablation and covered by the ablation zone in the target tumor and surrounding ablation margin using imaging criteria

IPD SHARING:
Plan to Share IPD: Undecided